CLINICAL TRIAL: NCT04855240
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ACP-044 for Acute Postoperative Pain Following Orthopedic Surgery (Bunionectomy)
Brief Title: Evaluate the Efficacy and Safety of ACP-044 for the Treatment of Acute Postoperative Pain Following Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-044-004
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Results first posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-02

CONDITIONS: Acute Postoperative Pain; Bunionectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Drug - ACP-044 Dose A (Experimental): ACP-044 Dose A
  Interventions: Drug: ACP-044 Dose A
- Drug - ACP-044 Dose B (Experimental): ACP-044 Dose B
  Interventions: Drug: ACP-044 Dose B
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACP-044 Dose A — Oral dose of ACP-044 Dose A
  Arms: Drug - ACP-044 Dose A
Drug: ACP-044 Dose B — Oral dose of ACP-044 Dose B
  Arms: Drug - ACP-044 Dose B
Drug: Placebo — Oral dose of placebo
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of ACP-044 compared with placebo in the treatment of acute postoperative pain

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and <60 years of age at the time of Screening
* Has a body mass index (BMI) <40 kg/m2
* Able to understand and provide signed informed consent
* Able to complete subject-reported outcome measures
* Is in need of a primary unilateral, first metatarsal bunionectomy with osteotomy and internal fixation under regional anesthesia and sedation
* Willing to remain inpatient at the study center for 4 days following surgery

Exclusion Criteria:

* Has had a contralateral foot bunionectomy in the past 3 months
* Has a planned concurrent surgical procedure (e.g. bilateral bunionectomy or collateral procedures like hammertoe correction on the surgical foot)
* Any subacute or chronic pain condition or use of a medication that would impair/impact the ability to rate the pain associated with the bunionectomy, in the opinion of the Investigator and Medical Monitor
* Has known or suspected regular use of opioids within the previous 6 months
* Has taken opioids within 24 hours prior to the scheduled surgery or within five half-lives of the drug, whichever is longer
* Has a known or suspected history of drug abuse, a positive drug screen at Screening or Day -1, or a recent (i.e., within the last 5 years) history of alcohol abuse. Subjects using marijuana are not allowed to participate in the study.
* Has taken any aspirin (ASA) or non-steroidal anti-inflammatory drugs (NSAIDs) within 2 days prior to the scheduled surgery or within five half-lives of the drug, whichever is longer
* Has initiated treatment with any medications within 1 month prior to study drug administration that could impact pain control or quantitation of their pain response
* Has been administered systemic steroids within five half-lives or 10 days prior to administration of study drug, whichever is longer
* Has current evidence, or medical history of a serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, endocrinologic, or other medical disorder, within the previous 12 weeks prior to Screening and on Day -1, that in the judgment of the Investigator and/or Medical Monitor would jeopardize the safe participation of the subject in the study. Also, subject must not have had a malignancy in the last year, with the exception of nonmetastatic basal cell of the skin or localized carcinoma in situ of the cervix.
* Is judged by the Investigator or the Medical Monitor to be inappropriate for the study

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Anaheim Clinical Trials, Anaheim, California
  - Chesapeake Ambulatory Surgery Center, Pasadena, Maryland
  - Endeavor Clinical Trials of San Antonio, TX, San Antonio, Texas
  - JBR Cinical Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug - ACP-044 400 mg Q6H: ACP-044 Dose A
  ACP-044 Dose A: Oral dose of ACP-044 400 mg Q6H
- Drug - ACP-044 1600 mg QD: ACP-044 Dose B
  ACP-044 Dose B: Oral dose of ACP-044 1600 mg QD
Period: Overall Study
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Started | 81 | 78 | 80
Completed | 77 | 73 | 75
Not Completed | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo | Total
Number analyzed (Participants) | 81 | 78 | 80 | 239
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (12.38) | 46.9 (10.93) | 42.7 (11.46) | 44.1 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 65 | 63 | 196
  Male | 13 | 13 | 17 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 26 | 22 | 70
  Not Hispanic or Latino | 58 | 52 | 58 | 168
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Primary Race: White | 62 | 58 | 58 | 178
  Primary Race: Black or African American | 16 | 14 | 17 | 47
  Primary Race: Asian | 3 | 2 | 3 | 8
  Primary Race: American Indian or Alaska Native | 0 | 3 | 0 | 3
  Primary Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Primary Race: Other | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 81 | 78 | 80 | 239

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of the Numeric Rating Scale (NRS) of Pain Intensity Scores From Time 0 (When First Dose on Day 1 is Administered) Through 24 Hours
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18, 21, and 24 hours.
Time Frame: 0-24 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Score on scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Score on scale * hour | 116.9 (5.55) | 129.0 (5.58) | 127.4 (5.52)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.1683, ANOVA; LSM difference = -10.5, 95% CI 2-sided [-25.4 to 4.4], Standard Error of Mean 7.61
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.8356, ANOVA; LSM difference = 1.6, 95% CI 2-sided [-13.4 to 16.6], Standard Error of Mean 7.64

2. Secondary Outcome: Time to First Rescue Medication Use After Time 0 (When First Dose on Day 1 is Administered)
Time Frame: 0-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
hours | 6.0 (0.5) | 5.7 (0.7) | 7.0 (0.7)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.2280, Log Rank; Hazard Ratio (HR) = 0.831, 95% CI 2-sided [0.598 to 1.155]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.5604, Log Rank; Hazard Ratio (HR) = 1.100, 95% CI 2-sided [0.793 to 1.527]

3. Secondary Outcome: Proportion of Subjects Who Were Opioid Free Through 24 Hours
Time Frame: 0-24 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Participants | 48 | 34 | 40
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.2457, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.11, 95% CI 2-sided [-0.05 to 0.26]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.3997, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.06, 95% CI 2-sided [-0.22 to 0.09]

4. Secondary Outcome: Proportion of Subjects Who Were Opioid Free Through 48 Hours
Time Frame: 0-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Participants | 45 | 32 | 40
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.4771, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.07, 95% CI 2-sided [-0.09 to 0.22]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.2925, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.09, 95% CI 2-sided [-0.24 to 0.06]

5. Secondary Outcome: Proportion of Subjects Who Were Opioid Free Through 72 Hours
Time Frame: 0-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Participants | 44 | 31 | 39
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.4628, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.07, 95% CI 2-sided [-0.09 to 0.22]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.3090, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.09, 95% CI 2-sided [-0.24 to 0.06]

6. Secondary Outcome: Mean AUC of the NRS of Pain Intensity Scores From Time 0 Through 48 Hours for ACP-044
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18, 21, 24, 30, 36, 42, and 48 hours.
Time Frame: 0-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Score on scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Score on scale * hour | 206.8 (11.21) | 229.7 (11.27) | 224.5 (11.12)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.2494, ANOVA; LSM difference = -17.7, 95% CI 2-sided [-47.8 to 12.4], Standard Error of Mean 15.36
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.7385, ANOVA; LSM difference = 5.1, 95% CI 2-sided [-25.1 to 35.4], Standard Error of Mean 15.42

7. Secondary Outcome: Mean AUC of the NRS of Pain Intensity Scores From Time 0 Through 72 Hours for ACP-044
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 15, 18, 21, 24, 30, 36, 42, 48, 54, 60, 66, and 72 hours.
Time Frame: 0-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Score on scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Score on scale * hour | 274.3 (16.72) | 304.7 (16.81) | 296.9 (16.59)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.3238, ANOVA; LSM difference = -22.6, 95% CI 2-sided [-67.5 to 22.3], Standard Error of Mean 22.91
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.7344, ANOVA; LSM difference = 7.8, 95% CI 2-sided [-37.3 to 52.9], Standard Error of Mean 22.99

8. Secondary Outcome: Mean AUC of the NRS of Pain Intensity Scores From Time 0 Through 4 Hours for ACP-044
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 0, 1, 2, 3, and 4 hours.
Time Frame: 0-4 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Score on scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Score on scale * hour | 18.3 (1.25) | 20.5 (1.26) | 18.6 (1.24)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.8489, ANOVA; LSM difference = -0.3, 95% CI 2-sided [-3.7 to 3.0], Standard Error of Mean 1.72
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.2768, ANOVA; LSM difference = 1.9, 95% CI 2-sided [-1.5 to 5.3], Standard Error of Mean 1.72

9. Secondary Outcome: Mean AUC of the NRS of Pain Intensity Scores From Time 0 Through 6 Hours for ACP-044
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 0, 1, 2, 3, 4, 5, and 6 hours.
Time Frame: 0-6 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Score on scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Score on scale * hour | 28.6 (1.86) | 32.4 (1.86) | 29.8 (1.84)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H; Test type: Superiority; p = 0.6291, ANOVA; LSM difference = -1.2, 95% CI 2-sided [-6.2 to 3.8], Standard Error of Mean 2.54
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.3182, ANOVA; LSM difference = 2.5, 95% CI 2-sided [-2.5 to 7.5], Standard Error of Mean 2.55

10. Secondary Outcome: Mean AUC of the NRS of Pain Intensity Scores From Time 0 Through 12 Hours for ACP-044
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 hours.
Time Frame: 0-12 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: Score on scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Score on scale * hour | 61.7 (3.18) | 66.6 (3.19) | 65.9 (3.15)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.3299, ANOVA; LSM difference = -4.2, 95% CI 2-sided [-12.8 to 4.3], Standard Error of Mean 4.35
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.8822, ANOVA; LSM difference = 0.6, 95% CI 2-sided [-7.9 to 9.2], Standard Error of Mean 4.37

11. Secondary Outcome: Mean AUC of the NRS of Pain Intensity Scores From 24 Through 48 Hours for ACP-044
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 24, 30, 36, 42, and 48 hours.
Time Frame: 24-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
score on a scale * hour | 90.2 (6.29) | 100.8 (6.32) | 97.3 (6.24)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.4094, ANOVA; LSM difference = -7.1, 95% CI 2-sided [-24.0 to 9.8], Standard Error of Mean 8.62
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.6901, ANOVA; LSM difference = 3.4, 95% CI 2-sided [-13.5 to 20.4], Standard Error of Mean 8.65

12. Secondary Outcome: Mean AUC of the NRS of Pain Intensity Scores From Time 48 Through 72 Hours for ACP-044
Description: Pain (efficacy) assessments were recorded hourly (±15 minutes) for a 12-hour interval on Day 1 beginning immediately prior to the fifth dose (time 0) administered in the study. Pain assessments were continued every 3 hours during the subsequent 12 hour interval, and then every 6 hours thereafter until 72 hours, then once daily in the morning until the follow-up clinical visit. Pain assessments were also obtained immediately prior to the administration of rescue medication.
  A 0 to 10 Numeric Rating Scale of Pain Intensity (NRS) was used to assess the subject's pain.
  Subjects were asked: "Please describe your foot pain at the present time from 0 to 10 where "0" means "no pain at all" and "10" means "the worst pain imaginable." The area under the curve is generated using the following timepoints beginning immediately prior to the fifth dose (time 0): 48, 54, 60, 66, and 72 hours.
Time Frame: 48-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale * hour
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
score on a scale * hour | 67.9 (6.27) | 75.4 (6.32) | 73.0 (6.22)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.5536, ANOVA; LSM difference = -5.1, 95% CI 2-sided [-21.9 to 11.7], Standard Error of Mean 8.59
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.7811, ANOVA; LSM difference = 2.4, 95% CI 2-sided [-14.5 to 19.3], Standard Error of Mean 8.64

13. Secondary Outcome: Rescue Medication Taken During 0-24 Hours
Description: Number of instances of rescue medication taken during first 24 hours.
Time Frame: 0-24 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: instances
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
instances | 2.1 (0.21) | 2.6 (0.21) | 2.3 (0.21)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.5267, ANOVA; LSM difference = -0.2, 95% CI 2-sided [-0.8 to 0.4], Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.3228, ANOVA; LSM difference = 0.3, 95% CI 2-sided [-0.3 to 0.9], Standard Error of Mean 0.29

14. Secondary Outcome: Rescue Medication Taken During 24-48 Hours
Description: Number of instances of rescue medication taken during 24-48 hours.
Time Frame: 24-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: instances
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
instances | 1.0 (0.17) | 1.2 (0.17) | 1.1 (0.17)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.7617, ANOVA; LSM difference = -0.1, 95% CI 2-sided [-0.5 to 0.4], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.6241, ANOVA; LSM difference = 0.1, 95% CI 2-sided [-0.4 to 0.6], Standard Error of Mean 0.24

15. Secondary Outcome: Rescue Medication Taken During 48-72 Hours
Description: Number of instances of rescue medication taken during 48-72 hours.
Time Frame: 48-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: instances
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
instances | 0.5 (0.12) | 0.7 (0.12) | 0.6 (0.12)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.3442, ANOVA; LSM difference = -0.2, 95% CI 2-sided [-0.5 to 0.2], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.7896, ANOVA; LSM difference = 0.0, 95% CI 2-sided [-0.3 to 0.4], Standard Error of Mean 0.17

16. Secondary Outcome: Rescue Medication Taken During 0-48 Hours
Description: Number of instances of rescue medication taken during first 48 hours.
Time Frame: 0-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: instances
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
instances | 3.1 (0.35) | 3.7 (0.35) | 3.3 (0.35)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.6003, ANOVA; LSM difference = -0.3, 95% CI 2-sided [-1.2 to 0.7], Standard Error of Mean 0.49
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.4086, ANOVA; LSM difference = 0.4, 95% CI 2-sided [-0.6 to 1.4], Standard Error of Mean 0.49

17. Secondary Outcome: Rescue Medication Taken During 0-72 Hours
Description: Number of instances of rescue medication taken during first 72 hours.
Time Frame: 0-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: instances
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
instances | 3.6 (0.43) | 4.4 (0.43) | 4.0 (0.43)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.4958, ANOVA; LSM difference = -0.4, 95% CI 2-sided [-1.6 to 0.8], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.4595, ANOVA; LSM difference = 0.5, 95% CI 2-sided [-0.8 to 1.7], Standard Error of Mean 0.61

18. Secondary Outcome: Proportion of Subjects Who Did Not Use Rescue Medication Through 24 Hours
Time Frame: 0-24 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 77 | 79
Participants | 16 | 10 | 10
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.1686, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.08, 95% CI 2-sided [-0.04 to 0.19]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.8333, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.10 to 0.11]

19. Secondary Outcome: Proportion of Subjects Who Did Not Use Rescue Medication Through 48 Hours
Time Frame: 0-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 77 | 79
Participants | 16 | 9 | 9
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.1939, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.02 to 0.20]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.9595, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.10 to 0.10]

20. Secondary Outcome: Proportion of Subjects Who Did Not Use Rescue Medication Through 72 Hours
Time Frame: 0-72 Hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 78 | 77 | 79
Participants | 16 | 9 | 9
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.1894, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.02 to 0.20]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.9595, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.10 to 0.10]

21. Secondary Outcome: Proportion of Subjects Who Are Pain Free (NRS ≤2) at 24 Hours
Time Frame: 0-24 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 78 | 76 | 75
Participants | 30 | 19 | 22
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.7117, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.06 to 0.24]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.7599, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.19 to 0.10]

22. Secondary Outcome: Proportion of Subjects Who Are Pain Free (NRS ≤2) at 48 Hours
Time Frame: 0-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 77 | 73 | 75
Participants | 42 | 37 | 41
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H; Test type: Superiority; p = 0.7070, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.00, 95% CI 2-sided [-0.16 to 0.16]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.6877, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.20 to 0.12]

23. Secondary Outcome: Proportion of Subjects Who Are Pain Free (NRS ≤2) at 72 Hours
Time Frame: 0-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 77 | 72 | 76
Participants | 50 | 49 | 55
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.8690, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.07, 95% CI 2-sided [-0.22 to 0.07]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.3790, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.19 to 0.10]

24. Secondary Outcome: Number of Hours Subjects Are Pain Free (NRS ≤2)
Time Frame: 0-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
hours | 29.0 (2.48) | 22.8 (2.49) | 23.0 (2.46)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.0897, ANOVA; LSM difference = 5.9, 95% CI 2-sided [-0.9 to 12.8], Standard Error of Mean 3.49
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.9434, ANOVA; LSM difference = -0.2, 95% CI 2-sided [-7.1 to 6.7], Standard Error of Mean 3.50

25. Secondary Outcome: Proportion of Subjects Who Were Opioid Free During 24-48 Hours
Time Frame: 24-48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Participants | 65 | 59 | 59
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.8355, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.09, 95% CI 2-sided [-0.04 to 0.21]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.3561, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.02, 95% CI 2-sided [-0.12 to 0.15]

26. Secondary Outcome: Proportion of Subjects Who Were Opioid Free During 48-72 Hours
Time Frame: 48-72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 79 | 78 | 80
Participants | 72 | 65 | 70
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.9413, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.06 to 0.13]
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.7819, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.04, 95% CI 2-sided [-0.15 to 0.07]

27. Secondary Outcome: Global Evaluation of Study Drug Just Before Time of First Rescue Medication Relative to Time 0 (When First Dose on Day 1 is Administered)
Description: 5 point scale (0-4) with categories of 0-poor, 1-fair, 2-good, 3-very good, or 4-excellent
Time Frame: First rescue medication dose, up to 24 hours post first dose.
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 59 | 61 | 61
score on a scale | 1.2 (0.16) | 1.5 (0.15) | 1.2 (0.15)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.8461, ANOVA; LSM difference = -0.0, 95% CI 2-sided [-0.5 to 0.4], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.1727, ANOVA; LSM difference = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.22

28. Secondary Outcome: Global Evaluation of Study Drug at the End of 24 Hours Relative to Time 0 (When First Dose on Day 1 is Administered)
Description: 5 point scale (0-4) with categories of 0-poor, 1-fair, 2-good, 3-very good, or 4-excellent
Time Frame: 24 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 67 | 62 | 66
score on a scale | 1.7 (0.16) | 2.0 (0.16) | 1.7 (0.16)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.9022, ANOVA; LSM difference = 0.0, 95% CI 2-sided [-0.4 to 0.5], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.2450, ANOVA; LSM difference = 0.3, 95% CI 2-sided [-0.2 to 0.7], Standard Error of Mean 0.23

29. Secondary Outcome: Global Evaluation of Study Drug at the End of 48 Hours Relative to Time 0 (When First Dose on Day 1 is Administered)
Description: 5 point scale (0-4) with categories of 0-poor, 1-fair, 2-good, 3-very good, or 4-excellent
Time Frame: 48 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 75 | 75 | 74
score on a scale | 2.2 (0.15) | 2.2 (0.15) | 2.0 (0.15)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.4205, ANOVA; LSM difference = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.4205
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.4336, ANOVA; LSM difference = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.21

30. Secondary Outcome: Global Evaluation of Study Drug at the End of 72 Hours Relative to Time 0 (When First Dose on Day 1 is Administered)
Description: 5 point scale (0-4) with categories of 0-poor, 1-fair, 2-good, 3-very good, or 4-excellent
Time Frame: 72 hours
Population: Two subjects in the ACP-044 Q6H group were included in the safety analysis set but not the full analysis set.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
Number analyzed (Participants) | 76 | 75 | 76
score on a scale | 2.3 (0.16) | 2.4 (0.16) | 2.1 (0.16)
Statistical Analysis 1: Comparison: Drug - ACP-044 400 mg Q6H vs Placebo; Test type: Superiority; p = 0.2718, ANOVA; LSM difference = 0.2, 95% CI 2-sided [-0.2 to 0.7], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Drug - ACP-044 1600 mg QD vs Placebo; Test type: Superiority; p = 0.1727, ANOVA; LSM difference = 0.3, 95% CI 2-sided [-0.1 to 0.7], Standard Error of Mean 0.22

ADVERSE EVENTS:
Time Frame: 62 days
Arm/Group | Drug - ACP-044 400 mg Q6H | Drug - ACP-044 1600 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/78 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/81 | 1/78 | 0/80
Other Adverse Events (participants affected / at risk) | 25/81 | 26/78 | 27/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug - ACP-044 400 mg Q6H (N=81) | Drug - ACP-044 1600 mg QD (N=78) | Placebo (N=80)
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0
acute pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Drug - ACP-044 400 mg Q6H (N=81) | Drug - ACP-044 1600 mg QD (N=78) | Placebo (N=80)
Nausea (Gastrointestinal disorders) | 15 | 10 | 11
Vomiting (Gastrointestinal disorders) | 5 | 7 | 3
Constipation (Gastrointestinal disorders) | 2 | 3 | 5
Headache (Nervous system disorders) | 10 | 13 | 13
Dizziness (Nervous system disorders) | 7 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT04855240/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT04855240/SAP_001.pdf